CLINICAL TRIAL: NCT03788395
Title: The Use of an Innovative Device for Therapeutic Adherence in Pediatric Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Coordinator of the group "Clinical and Environmental Epidemiology of Pulmonary and Allergic Pediatric Diseases". Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/2018
Record Dates: First submitted 2018-12-21; First posted 2018-12-27 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symbicort Turbohaler plus Turbo+ (Experimental): 10 asthmatic children
  Interventions: Device: Symbicort Turbohaler plus Turbo+
- Symbicort Turbohaler without Turbo+ (Active Comparator): 10 asthmatic children
  Interventions: Drug: Symbicort Turbohaler without Turbo+

INTERVENTIONS:
Device: Symbicort Turbohaler plus Turbo+ — Symbicort Turbohaler (Budesonide and Formoterol Fumarate Dihydrate) plus Turbo+ for three months.
  Arms: Symbicort Turbohaler plus Turbo+
Drug: Symbicort Turbohaler without Turbo+ — Symbicort Turbohaler (Budesonide and Formoterol Fumarate Dihydrate) without Turbo+ for three months.
  Arms: Symbicort Turbohaler without Turbo+

SUMMARY:
The management of chronic diseases requires a constant monitoring of treatment adherence, in order to obtain an optimal disease control. However, this is often difficult to achieve, especially in pediatric age.

In this sense, for asthmatic patients treated by Symbicort Turbohaler, "AstraZeneca" developed the "Turbo+", an electronic device attached to the Turbohaler, which allows to feel whether the patient does the inhalation, and to register it on a specific application.

The present randomized trial aims to compare the treatment adherence between asthmatic children/adolescents aged 6-17 years treated with Symbicort Turbohaler plus Turbo+ or Symbicort Turbohaler without Turbo+.

ELIGIBILITY:
Inclusion Criteria:

- uncontrolled mild or moderate persistent asthma;

Exclusion Criteria:

* acute upper respiratory infections;
* immunological or metabolic systemic disease;
* major malformations of the upper airways;
* active smokers.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Rating Scale (MARS) | 3 months
  Change in the MARS score from baseline to the end of treatment

SECONDARY OUTCOMES:
Childhood Asthma Control Test (C-ACT) | 3 months
  Change in the C-ACT score from baseline to the end of treatment
Asthma Control Test (ACT) | 3 months
  Change in the ACT score from baseline to the end of treatment
Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | 3 months
  Change in the PAQLQ score from baseline to the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614